CLINICAL TRIAL: NCT02900508
Title: Virtual Reality-based Training in Cerebellar Ataxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201410010A
Record Dates: First submitted 2016-09-06; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Cerebellar Ataxia
MeSH Terms: conditions — Cerebellar Ataxia

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Exergaming training (Experimental): Participants in the exergaming training group received a 4-week exergaming intervention.
  Interventions: Other: Exergaming training
- Control training (Active Comparator): Participants in the control training group received a 4-week conventional training.
  Interventions: Other: Physical therapy intervention

INTERVENTIONS:
Other: Exergaming training
  Arms: Exergaming training
Other: Physical therapy intervention
  Arms: Control training

SUMMARY:
The purpose of this study was to investigate the effects of virtual reality-base training for cerebellar ataxia.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of SCA 1, 2, 3 and 6 by a neurologist
* ability to walk independently with or without any walking aids
* age ≥ 20
* a score of ≥ 24 on the mini-mental state examination

Exclusion Criteria:

* histories of other neurological, cardiovascular, or orthopedic diseases affecting motor performance and balance
* uncontrolled chronic diseases

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Scale for the Assessment and Rating of Ataxia | Change from baseline at 4 weeks
Alternate nose to finger test | Change from baseline at 4 weeks
Alternate heel on shin test | Change from baseline at 4 weeks

SECONDARY OUTCOMES:
Nine-hole peg test | Change from baseline at 4 weeks
Walking speed | Change from baseline at 4 weeks
Step width | Change from baseline at 4 weeks